CLINICAL TRIAL: NCT02661243
Title: Implantology and Sjögren's Syndrome: a Multicenter Prospective Cohort Study
Brief Title: Implantology and Sjögren's Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derk Jan Jager (Other)
Collaborators: UMC Utrecht (Other); University Medical Center Groningen (Other); Tandartspraktijk Bocht Oosterdiep (Unknown); Isala (Other); BioHorizons, Inc. (Industry); Fonds NutsOhra (Other)
Responsible Party: Sponsor-Investigator, Derk Jan Jager, PhD, Amsterdam UMC, location VUmc
Organization: Amsterdam UMC, location VUmc (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL47808.029.14
Record Dates: First submitted 2016-01-18; First posted 2016-01-22 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Sjogren's Syndrome
Keywords: Sjogren's Syndrome; Dental Implants
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Dentate Sjogren's syndrome arm (Other): 30 human adults affected by SS with the need of replacement of missing premolars or molars in the upper or lower jaw. Intervention: insertion of Biohorizons Laser-lok bonelevel dental implants
  Interventions: Device: Biohorizons Laser-lok bonelevel dental implants
- Dentate healthy controls arm (Other): 30 healthy human adults with the need of replacement of missing premolars or molars in the upper or lower jaw. Intervention: insertion of Biohorizons Laser-lok bonelevel dental implants
  Interventions: Device: Biohorizons Laser-lok bonelevel dental implants
- Edentulous Sjogren's syndrome arm (Other): 30 human edentulous adults affected by SS with the need of stabilization of the dentures. Intervention: insertion of Biohorizons Laser-lok bonelevel dental implants
  Interventions: Device: Biohorizons Laser-lok bonelevel dental implants
- Edentulous healthy controls arm (Other): 30 healthy human edentulous adults with the need of stabilization of the dentures. Intervention: insertion of Biohorizons Laser-lok bonelevel dental implants
  Interventions: Device: Biohorizons Laser-lok bonelevel dental implants

INTERVENTIONS:
Device: Biohorizons Laser-lok bonelevel dental implants — Insertion of Biohorizons Laser-lok bonelevel dental implants to replace missing (pre)molars or to stabilize a denture

SUMMARY:
Until now it has not been investigated whether placement of implants in SS patients is less successful than compared to non-SS patients. The risk factors and the efficacy of dental implants in dry mouth patients are not known because of the lack of scientific evidence. The aim of this study is to investigate changes in marginal peri-implant bone loss and the clinical performance of dental implants in SS patients compared to implants in healthy patients.

DETAILED DESCRIPTION:
Rationale: Until now it has not been investigated whether placement of implants in SS patients is less successful than compared to non-SS patients. The risk factors and the efficacy of dental implants in dry mouth patients are not known because of the lack of scientific evidence.

Objective: to investigate changes in marginal peri-implant bone loss and the clinical performance of dental implants in SS patients compared to implants in healthy patients.

Study design: A prospective multicenter clinical trial.

Study population: N = 120

Intervention: All patients receive Biohorizons Laser-lok bonelevel implants to replace the missing (pre)molars or to support a full denture in the upper and lower jaw .

This study is comprised of four study groups:

* 30 human adults affected by SS with the need of replacement of missing premolars or molars in the upper or lower jaw.
* 30 healthy human adults with the need of replacement of missing premolars or molars in the upper or lower jaw.
* 30 human edentulous adults affected by SS with the need of stabilization of the dentures.
* 30 healthy human edentulous adults with the need of stabilization of the dentures.

Main study parameters/endpoints: changes in marginal peri-implant bone loss of dental implants between the healthy and SS groups and differences in clinical performance 1.5 years after finalization.

ELIGIBILITY:
Inclusion criteria (dentate group, Sjögren):

* The patient is at least 18 years and younger than 70;
* A diagnosed (by the AECG guidelines; see attachment; Vitali et al., 2002) primary or secondary Syndrome of Sjögren;
* The missing or lost tooth/teeth are premolars and/or molars in the upper or lower jaw.
* Sufficient healthy and vital bone to insert a dental implant with a minimum length of 8 mm and at least 3.8 mm in diameter. In case of insufficient bone volume, a bone augmentation procedure will be performed with autologue bone. If necessary the autologue bone can be mixed with artificial bone (artificial bone graft substitutes in combination with a membrane).
* The implant site must be free from infection;
* Adequate oral hygiene (modified plaque index and modified sulcus bleeding index ≤ 1) (Mombelli et al., 1987; Loe and Silness, 1963)
* Sufficient mesio-distal, bucco-lingual, and interocclusal space for placement of an anatomic restoration;
* The patient is capable of understanding and giving informed consent.

Inclusion criteria (edentulous group, Sjögren):

* The patient is at least 18 years and younger than 70;
* A diagnosed (by the AECG guidelines; Vitali et al., 2002) primary or secondary Syndrome of Sjögren
* The patient is edentulous. Before final inclusion in the study the patient has to be edentulous for 1 year.
* Problems with conventional denture retention, stability and/or adaptation, which could be solved by an implant, supported denture (lower or/and upper jaw).
* Sufficient healthy and vital bone to insert dental implants with a minimum length of 8 mm and at least 3.8 mm in diameter. In case of insufficient bone volume, a bone augmentation procedure will be performed with autologue bone. If necessary the autologue bone can be mixed with artificial bone (artificial bone graft substitutes in combination with a membrane).
* The implant site must be free from infection;
* Capable of performing adequate oral hygiene;
* The patient is capable of understanding and giving informed consent.

Inclusion criteria control groups:

- The inclusion criteria for the healthy control groups are similar as for the Sjögren groups without the Sjögren criterion.

Exclusion criteria:

Criteria used for excluding patients from this study are as follows:

* Medical and general contraindications for the surgical procedures;
* Presence of an active and uncontrolled periodontal disease as expressed by probing pockets depths > 4mm with bleeding upon probing;
* Smoking (patients who stop smoking six weeks before the operation can be included);
* A history of radiotherapy to the head and neck region;
* Use of intravenous bisphosphonates or the use of oral bisphosphonates for more than 5 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2015-05; Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Change in marginal peri-implant bone loss of dental implants | 1.5 years
  changes in marginal peri-implant bone loss of dental implants between the healthy and SS groups and differences in clinical performance 1.5 years after finalization.

SECONDARY OUTCOMES:
Implant survival | 1.5 years
  The survival rate of the fixture is assessed 1 month, 6 months, 1 year and 1.5 years after placement of the definitive restoration. Implant survival is defined as presence of the implant at time of the follow-up examinations.
Overdenture/crown survival | 1.5 years
  The survival (i.e. fully intact) rate of the denture or crown is assessed 1 month, 6 months, 1 year and 1.5 years after placement of the definitive restoration.
Modified Plaque-index and Modified Bleeding-Index | 1.5 years
  These parameters are evaluated pre-operative, 1 month, 6 months, 1 year and 1.5 years after placement of the definitive restoration. The adjacent teeth are counted as well in the assessments (dentate groups only).
Probing depth | 1.5 years
  Probing of the implant and the adjacent teeth (dentate groups only) is performed at three sites, buccodistal, buccomedial, buccomesial. The probing depth is measured 1 month, 6 months, one year and 1.5 years after placement of the definitive restoration.
Width of keratinized epithelium | 1.5 years
  The width in millimetres of keratinized epithelium is measured pre-operative, 1 month, 6 months, 1 year and 1.5 years after the definitive restoration has been placed. For this a periodontal probe is used.
Patient satisfaction and impact of oral health on the quality of life | 1.5 years
  - All patients: OHIP-NL14. Oral Health Impact Profile. An instrument for measuring the impact of oral health on the quality of life. A validated Dutch-language version of the OHIP-14, a questionnaire by means of which the impact of oral health on the quality of life of patients can be determined is completed by every participant at every examination
Denture function and satisfaction | 1.5 years
  * Edentulous groups: the following validated questionnaires are used for the edentulous groups only (see attachment; Vervoorn et al., 1988):
  * A. General experience with the denture, including a grade from 1 tot 10
  * B. Complaints form with regard to aesthetics and function of the denture
  * C. Chewing list (which food can be chewed well and which food is difficult to chew).
  The participant at every time point completes these questionnaires
Disease symptoms (SS groups only) | 1.5 years
  patients in the SS groups are asked to complete the EULAR Sjögren's Syndrome Patient Reported Index and the EULAR Sjögren's Syndrome Disease Activity Index (ESSPRI & ESSDAI; see attachment) questionnaire with regard to disease symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Derk Jan Jager, DMD, PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (5):
- Netherlands (5):
  - VU Medical Center department of Maxillofacial surgery, Amsterdam
  - University Medical Center Groningen, Groningen
  - University Medical Center Utrecht, Utrecht
  - Tandartspraktijk Bocht Oosterdiep, Veendam
  - Vogellanden Center for Special Care Dentistry/Isala, Zwolle

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] den Hartog L, Slater JJ, Vissink A, Meijer HJ, Raghoebar GM. Treatment outcome of immediate, early and conventional single-tooth implants in the aesthetic zone: a systematic review to survival, bone level, soft-tissue, aesthetics and patient satisfaction. J Clin Periodontol. 2008 Dec;35(12):1073-86. doi: 10.1111/j.1600-051X.2008.01330.x. PMID 19040585
- [Background] Pecora GE, Ceccarelli R, Bonelli M, Alexander H, Ricci JL. Clinical evaluation of laser microtexturing for soft tissue and bone attachment to dental implants. Implant Dent. 2009 Feb;18(1):57-66. doi: 10.1097/ID.0b013e31818c5a6d. PMID 19212238
- [Background] Fox RI. Sjogren's syndrome. Lancet. 2005 Jul 23-29;366(9482):321-31. doi: 10.1016/S0140-6736(05)66990-5. PMID 16039337
- [Background] Vitali C, Bombardieri S, Jonsson R, Moutsopoulos HM, Alexander EL, Carsons SE, Daniels TE, Fox PC, Fox RI, Kassan SS, Pillemer SR, Talal N, Weisman MH; European Study Group on Classification Criteria for Sjogren's Syndrome. Classification criteria for Sjogren's syndrome: a revised version of the European criteria proposed by the American-European Consensus Group. Ann Rheum Dis. 2002 Jun;61(6):554-8. doi: 10.1136/ard.61.6.554. PMID 12006334
- [Background] Meijndert L, Meijer HJ, Raghoebar GM, Vissink A. A technique for standardized evaluation of soft and hard peri-implant tissues in partially edentulous patients. J Periodontol. 2004 May;75(5):646-51. doi: 10.1902/jop.2004.75.5.646. PMID 15212345